CLINICAL TRIAL: NCT01387581
Title: To Excise or Not?: Comparing Clinical Management Decisions for Melanoma Between Dermatologists With and Without the Aid of MelaFind
Brief Title: Does the Aid of MelaFind Affect Clinical Management Decisions
Status: Completed | Type: Observational
Sponsor: MELA Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20101
Record Dates: First submitted 2011-06-28; First posted 2011-07-04 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Without MelaFind: Study dermatologists will review clinical exam information and 3 high quality digital images for each lesion without MelaFind result.
- With MelaFind: Study dermatologists will review clinical exam information, 3 high quality digital images, and MelaFind result for each lesion
- Experts Without MelaFind: PSL Experts, prospectively identified and recruited by the PI after the general recruitment is completed. They will review clinical exam information and 3 high quality digital images for each lesion without MelaFind result.

SUMMARY:
The objective of this study is to determine and compare the performance of dermatologists (in Germany) on the excision decision against the performance of MelaFind, a non-invasive and objective multi-spectral computer vision system designed as a tool to aid dermatologists in the detection of early melanoma. The hypothesis is that MelaFind's sensitivity is superior to the average excisions sensitivity of dermatologists.

Another objective is to determine and compare the performance of dermatologists (in Germany) with and without the aid of MelaFind. The hypothesis is that the average excision sensitivity of dermatologists with the aid of MelaFind is superior to the average excision sensitivity of dermatologists without the aid of MelaFind.

A similar study was previously conducted with dermatologists in the US (NCT01011153). An exploratory objective is to compare the excision decisions of dermatologists from the previous study (in the US) to dermatologists in in this study (in Germany).

DETAILED DESCRIPTION:
Early detection of melanoma is critical for favorable prognosis, since patients with earlier stage melanomas have a much higher probability of survival than with later stages. The traditional method of early detection has been with serial total body skin exams where the health care provider examines all skin surfaces, including mucosa, for suspicious pigmented lesions. The diagnostic performance of dermatologists for melanoma depends on the level of dermatological training. More important than being able to make a diagnosis of melanoma on clinical impression is the ability to make an appropriate decision to excise the lesion. To aid dermatologists in the detection of early melanoma, MelaFind was developed, a non-invasive and objective multi-spectral computer vision system technology. It was designed to generate output - MelaFind Positive or MelaFind Negative- for consideration in the lesion management decisions.

This survey study will determine and compare the average excision sensitivity to melanoma and specificity of dermatologists (in Germany) without MelaFind output to the average excision sensitivity to melanoma and specificity of dermatologists (in Germany) with MelaFind output. Another purpose is to determine and compare the sensitivity to melanoma and specificity of MelaFind to the average excision sensitivity to melanoma and specificity of dermatologists without MelaFind output.

ELIGIBILITY:
Inclusion Criteria:

-Only board certified dermatologists

Exclusion Criteria:

-May not have previously participated in MELA Protocols 20061, 20081 or 20063

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 130 dermatologists will enter by way of general invitation and will be randomly placed in either Arm 1 (Without MelaFind) or Arm 2 (With MelaFind). Another group, up to 30 Pigmented Skin Lesion Experts, will be prospectively identified by the Principal Investigator of this study prior to any participant recruitment, and will be invited to participate in the study by the PI after the general recruitment is completed.
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Hauschild, MD, Principal Investigator — Dermatologic Cooperative Oncology Group
Locations (1):
- MELA Sciences, Irvington, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dermatologists were selected at random from Germany's public dermatology membership list and were invited to participate by letter. Those interested in participating were asked to register online. Eligible dermatologists were selected to participate on a first-come basis and were divided by random placement into one of two study arms.
Pre-assignment Details: Dermatologists interested in participating were asked to register online by responding to an Intake Survey. The survey included questions about dermatology training, medical licensure, board certification, and comfort with and frequency of screening for melanoma. Only board certified dermatologists were permitted to participate in the study.
Period: Overall Study
Arm/Group | Without MelaFind | With MelaFind | Experts Without MelaFind
Started | 108 | 107 | 12
Completed | 101 | 101 | 9
Not Completed | 7 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Without MelaFind | With MelaFind | Experts Without MelaFind | Total
Number analyzed (Participants) | 101 | 101 | 9 | 211
Age, Customized [Number; unit: participants]
  31-40 years | 18 | 22 | 2 | 42
  41-50 years | 48 | 44 | 5 | 97
  51-60 years | 29 | 30 | 2 | 61
  > 60 years | 6 | 5 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 1 | 85
  Male | 60 | 58 | 8 | 126
Region of Enrollment [Number; unit: participants]
  Germany | 101 | 101 | 9 | 211
Dermoscopy use [Number; unit: participants]
  Never | 0 | 0 | 0 | 0
  Rarely | 0 | 0 | 0 | 0
  < half of pigmented skin lesions | 4 | 16 | 3 | 23
  > half of pigmented skin lesions | 17 | 16 | 2 | 35
  Almost all | 28 | 31 | 1 | 60
  Always | 52 | 38 | 3 | 93
Years in Practice [Number; unit: participants]
  < 5 years | 1 | 0 | 0 | 1
  5 - 10 years | 8 | 17 | 1 | 26
  11 - 15 years | 26 | 23 | 2 | 51
  16 - 20 years | 27 | 25 | 4 | 56
  > 60 years | 39 | 36 | 2 | 77

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: Dermatologist sensitivity is the percent of melanomas that dermatologists selected to biopsy. MelaFind sensitivity is the percent of melanomas that MelaFind called "Positive."
Time Frame: Within 120 days of Data Lock
Measure: Mean (95% Confidence Interval); unit: percent of true positives
Arm/Group | Without MelaFind | With MelaFind | Experts Without MelaFind
Number analyzed (Participants) | 101 | 101 | 9
percent of true positives | 69.5 [64.3 to 76.0] | 78.0 [73.9 to 83.5] | 71.8 [66.3 to 77.9]

2. Primary Outcome: Specificity
Description: Dermatologist specificity is the percent of non-melanomas that dermatologists selected not to biopsy. MelaFind specificity is the percent of non-melanomas that MelaFind called "Negative."
Time Frame: Within 120 days of Data Lock
Measure: Mean (95% Confidence Interval); unit: percent of true negatives
Arm/Group | Without MelaFind | With MelaFind | Experts Without MelaFind
Number analyzed (Participants) | 101 | 101 | 9
percent of true negatives | 55.9 [47.3 to 60.5] | 45.8 [38.1 to 50.8] | 54.6 [46.3 to 59.7]

ADVERSE EVENTS:
Arm/Group | Without MelaFind | With MelaFind | Experts Without MelaFind
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/107 | 0/12
Other Adverse Events (participants affected / at risk) | 0/108 | 0/107 | 0/12

LIMITATIONS AND CAVEATS:
A limitation of this study is the reader study format. Lesions were presented to participating dermatologists as photographs via the online system. This presentation can only approximate an in-person clinical exam.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No